CLINICAL TRIAL: NCT00049127
Title: Phase I/II Trial of Imatinib Mesylate; (Gleevec; STI571) in Treatment of Recurrent Oligodendroglioma and Mixed Oligoastrocytoma
Brief Title: Imatinib Mesylate in Treating Patients With Recurrent Brain Tumor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N0272; NCI-2011-01576 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCCTG-N0272; CDR0000257812 (Registry Identifier: NCI Physician Data Query); U10CA025224 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Adult Anaplastic Oligodendroglioma; Adult Mixed Glioma; Adult Oligodendroglioma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Oligodendroglioma; Glioma; Brain Neoplasms | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase II (Group 1) (Experimental): Patients receive imatinib mesylate PO, at the MTD determined in phase I, BID for 4 weeks.
  Interventions: Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Phase II (Group 2) (Experimental): Patients receive standard-dose imatinib mesylate PO BID for 4 weeks.
  Interventions: Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP57148B; Gleevec; Glivec; STI 571; STI-571; STI571
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Pharmacological Study — Optional correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of imatinib mesylate and to see how well it works in treating patients with a recurrent brain tumor that has not responded to previous surgery and radiation therapy. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the maximum tolerated dose of imatinib (imatinib mesylate) in patients with recurrent oligodendroglioma and mixed oligoastrocytoma that are currently on enzyme inducing anticonvulsant therapy. (Study 1) II. To assess the efficacy of imatinib in patients with recurrent oligodendrogliomas and mixed oligoastrocytomas (with pathologic evidence of oligodendrogliomatous component) as measured by progression-free survival, response, and overall survival. (Study 2) III. To acquire pilot data on a patient group not traditionally eligible for recurrent oligodendroglioma and mixed oligoastrocytoma clinical trials (those having > 2 prior chemotherapy regimens or 2 prior chemotherapy regimens for recurrent/progressive disease). (Study 3) IV. To examine the toxicity and safety of imatinib in patients with recurrent oligodendrogliomas and mixed oligoastrocytomas (with pathologic evidence of oligodendrogliomatous component). (Studies 1, 2, and 3) V. To perform a preliminary correlative study of 1p/19q alterations, alpha platelet-derived growth factor receptor (PDFGR) gene amplification and levels of related downstream signaling elements in tumor tissue, with clinical study endpoints. (Studies 1, 2, and 3) VI. To perform a descriptive correlative analysis of steady state pharmacokinetic data regarding imatinib and active metabolites with the study endpoints. (Studies 1, 2, and 3)

OUTLINE: This is a phase I, dose-escalation study followed by a phase II and a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Study 1 Arm C:

  * Currently on anticonvulsants which can induce cytochrome p450 (phenytoin, carbamazepine, barbiturates, primidone and if unsure contact study chair)
  * =< 2 prior chemotherapy regimens (with maximum of 1 prior chemotherapy regimen for recurrent disease)
* Study 2 Arms A and B:

  * On or off anticonvulsants
  * =< 2 prior chemotherapy regimens (with maximum of 1 prior chemotherapy regimen for recurrent disease)
* Study 3 Arms D and E:

  * On or off anticonvulsants
  * > 2 chemotherapy regimens or 2 prior chemotherapy regimens for progressive/recurrent disease
* All Arms:
* Histological confirmation of a grade 2-4 oligodendroglioma, or mixed oligoastrocytoma grade 2-4 containing oligodendrogliomatous component on central pathology review prior to study registration, and a diagnosis of recurrence; tissues from all available prior surgeries should be sent, in particular those from time of initial diagnosis
* Measurable or evaluable disease by magnetic resonance imaging (MRI) or computed tomography (CT) scan
* Fixed dose of corticosteroids (or no corticosteroids) for at least 1 week prior to the pre-study baseline scan
* Patients undergoing surgery for initial or progressive disease, must be at least 2 weeks from the date of surgery, must have recovered from the effects of their surgery, and must have unequivocal tumor growth on the pre-study baseline neuroimaging study as compared to the first post-operative scan, unless there is a separate lesion or residual disease compatible with tumor that is not within the surgical bed
* Unequivocal evidence of tumor progression by MRI or CT scan performed =< 21days prior to study registration
* Must have failed surgery/radiotherapy (RT) and Temozolomide or nitrosourea based therapy
* >= 12 weeks since the completion of RT
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets (PLT) >= 100,000/mm^3
* Hemoglobin (Hgb) >= 9 g/dL
* Total bilirubin =< 1.5 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x upper limit of normal (ULN)
* Creatinine =< 2.0 mg/dL
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
* >= 6 weeks since the last day of nitrosourea-based chemotherapy prior to study entry
* >= 4 weeks from any investigational agents prior to study entry
* >= 4 weeks from other chemotherapy prior to study entry
* >= 2 weeks from vincristine and biologic non-cytotoxic agents, e.g., tamoxifen, thalidomide, cis-retinoic acid, interferon, etc, prior to study entry
* Patients or designated individual(s) with durable medical power of attorney for the patient must be able to provide informed, written consent, and complete any required study questionnaire(s) within the specifications of this study

Exclusion Criteria:

* All Arms
* Receiving warfarin or heparin
* Received prior stereotactic radiosurgery, interstitial brachytherapy, or interstitial chemotherapy including carmustine (BCNU) wafers unless there is a separate lesion on MRI, which is not part of the previous treatment field
* Active uncontrolled infection
* History of myocardial infarction =< 6 months or congestive heart failure (CHF) requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias; patients must have a New York Heart Association (NYHA) of class II or less; (NYHA class I: patients with no limitation of activities; they suffer no symptoms from ordinary activities; class II: patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion; class III: patients with marked limitation of activity; they are comfortable only at rest; class IV: patients who should be at complete rest, confined to bed or chair; any physical activity brings on discomfort and symptoms occur at rest)
* Other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the interpretation of potential drug-induced toxicities
* Women of child-bearing potential, pregnant or nursing; such patients must have a negative pregnancy test (b-HCG) =< 7 days prior to study registration
* Men or women of childbearing potential, not willing to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.); the efficacy of oral contraceptives may be decreased in patients who receive p450-inducing anticonvulsants; for these patients, use of a second mode of contraception is recommended; patients of childbearing potential must utilize effective contraception and avoid becoming pregnant or fathering a child for 6 months after completing study drug
* Other active malignancy, besides skin carcinomas (must not be melanoma)
* Concomitant serious immunocompromised status (other than that related to concomitant steroids); patients that are human immunodeficiency virus (HIV) positive are eligible, provided that there is no other reason for exclusion, based on the eligibility as outlined elsewhere in this section
* Significant intratumoral hemorrhage on baseline MRI or CT, or other history of significant intratumoral hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-06 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Jaeckle, MD, Study Chair — Mayo
Locations (228):
- United States (228):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Rush - Copley Medical Center, Aurora, Illinois
  - Bromenn Lifecare Center, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Sarah Culbertson Memorial Hospital, Rushville, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Memorial Hospital, Onawa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Memorial Hospital of Arkansas City, Arkansas City, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Ottawa, Ottawa, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Center for Hematology- Oncology of Southern Michigan PLC, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Brainerd Medical Center Inc, Brainerd, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro-Minnesota NCI Community Oncology Research Program, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Adult and Pediatric Urology PLLP, Sartell, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine of Bozeman, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Fremont Area Medical Center, Fremont, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Bryan LGH Medical Center East, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Cancer Consortium-Upstate NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Cole, Sharon, K. M.D. (UIA Investigator), Kenton, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Stark, Michael, Edward. M.D. (UIA Investigator), Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Medical Center Clinic-Butler Office, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Sharon Regional Cancer Center, Hermitage, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical Center Clinic-Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford NCI Community Oncology Research Program of the North Central Plains, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Study 1 Arm C: Phase I patients on enzyme-inducing anticonvulsants (EIACs) and <=2 prior regimens
  Imatinib at assigned dose. Escalation of cohorts-of-3 per section 7.1 of the protocol. Assigned dose will be administered p.o. twice daily in divided doses.
- Study 2 Arm A: Phase II patients on enzyme-inducing anticonvulsants (EIACs) and <=2 prior regimens
  Imatinib at Maximum Tolerated Dose (MTD) from Study 1 mg p.o. bid daily
- Study 2 Arm B: Phase II patients not on enzyme-inducing anticonvulsants (EIACs) and <=2 prior regimens
  Imatinib at 300 mg b.i.d.
- Study 3 Arm D: Phase II patients on enzyme-inducing anticonvulsants (EIACs) and >2 prior regimens
  Imatinib at Maximum Tolerated Dose (MTD) from Study 1 mg p.o. bid daily
- Study 3 Arm E: Phase II patients not on enzyme-inducing anticonvulsants (EIACs) and >2 prior regimens
  Imatinib at 300 mg b.i.d.
Period: Overall Study
Arm/Group | Study 1 Arm C | Study 2 Arm A | Study 2 Arm B | Study 3 Arm D | Study 3 Arm E
Started | 12 | 0 | 40 | 0 | 12
Completed | 12 | 0 | 39 | 0 | 12
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study 1 Arm C: Phase I patients on EIACs and <=2 prior regimens
- Study 2 Arm A: Phase II patients on EIACs and <=2 prior regimens
- Study 2 Arm B: Phase II patients not on EIACs and <=2 prior regimens
- Study 3 Arm D: Phase II patients on EIACs and >2 prior regimens
- Study 3 Arm E: Phase II patients not on EIACs and >2 prior regimens
- Total: Total of all reporting groups
Arm/Group | Study 1 Arm C | Study 2 Arm A | Study 2 Arm B | Study 3 Arm D | Study 3 Arm E | Total
Number analyzed (Participants) | 12 | 0 | 39 | 0 | 12 | 63
Age, Continuous [Median (Full Range); unit: years]
  participants | 45 [34 to 65] |  | 46 [22 to 83] |  | 47 [22 to 59] | 46 [22 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 17 |  | 4 | 22
  Male | 11 |  | 22 |  | 8 | 41
Performance Score [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) PERFORMANCE STATUS:
  * 0=Asymptomatic and fully active
  * 1=Symptomatic; fully ambulatory; restricted in physically strenuous activity
  * 2=Symptomatic; ambulatory; capable of self-care; more than 50% of waking hours are spent out of bed
  * 3=Symptomatic; limited self-care; spends more than 50% of time in bed, but not bedridden
  * 4=Completely disabled; no self-care; bedridden
  participants
    0 | 7 |  | 10 |  | 6 | 23
    1 | 4 |  | 23 |  | 4 | 31
    2 | 1 |  | 6 |  | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival (PFS), Defined as a Patient Being Alive and Progression-free 183 Days After the Date of Registration.
Description: The proportion of successes will be estimated using the Binomial point estimator (number of successes divided by the total number of evaluable patients) and the Binomial 90% confidence interval estimated using the Duffy-Santer algorithm.
  Progression is defined using response criteria (the neurologic examination and the MRI and/or CT), >25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions.
Time Frame: 6 months
Measure: Number; unit: percentage of patients
Arm/Group | Study 1 Arm C | Study 2 Arm A | Study 2 Arm B | Study 3 Arm D | Study 3 Arm E
Number analyzed (Participants) | 12 | 0 | 39 | 0 | 12
percentage of patients | 33.35 |  | 33.3 |  | 25

2. Secondary Outcome: Confirmed Response (i.e., an Objective Status of Complete Response (CR), Partial Response (PR), or Regression (REGR) on 2 Successive Evaluations at Least 4 Weeks Apart After the Start of Study Treatment).
Description: Complete Response (CR) is defined using response criteria (the neurologic examination and the Magnetic resonance imaging (MRI) and/or Computerized Tomography (CT)), total disappearance of all tumor with patient off corticosteroids or only on adrenal replacement maintenance.
  Partial Response (PR) is defined using response criteria (the neurologic examination and the MRI and/or CT), >=50% reduction in product of perpendicular diameters of contrast enhancement or mass with no new lesions with the patient being on stable or decreased steroid dose.
  Regression (REGR) is defined using response criteria (the neurologic examination and the MRI and/or CT), unequivocal reduction in size of contrast-enhancement or decrease in mass effect as agreed upon independently by primary physician and quality control physicians; no new lesions. Patient should be on stable or decreased steroid dose.
Time Frame: Up to 5 years
Measure: Number; unit: percentage of confirmed responses
Arm/Group | Study 1 Arm C | Study 2 Arm A | Study 2 Arm B | Study 3 Arm D | Study 3 Arm E
Number analyzed (Participants) | 12 | 0 | 39 | 0 | 12
percentage of confirmed responses | 0 |  | 5.1 |  | 0

3. Secondary Outcome: Percentage of Patients Progression-free
Description: The percentage of patient progression-free at 12 months, 18 months, and PFS will be estimated. Kaplan-Meier survival curves and logrank tests will be used to estimate progression-time distributions.
  Progression is defined using response criteria (the neurologic examination and the MRI and/or CT), >25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions.
Time Frame: Time from study registration to date of disease progression or last follow-up, assessed up to 5 years
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Study 1 Arm C | Study 2 Arm A | Study 2 Arm B | Study 3 Arm D | Study 3 Arm E
Number analyzed (Participants) | 12 | 0 | 39 | 0 | 12
months | 1.9 [1.7 to NA] — Upper Confidence Interval (CI) was not reached |  | 4.0 [1.9 to 6.2] |  | 4.5 [2.2 to NA] — Upper CI was not reached

4. Secondary Outcome: Overall Time to Death
Description: Kaplan-Meier survival curves and logrank tests will be used to estimate survival distributions.
Time Frame: Time from date of registration to date of death due to any cause or last follow-up, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Study 1 Arm C | Study 2 Arm A | Study 2 Arm B | Study 3 Arm D | Study 3 Arm E
Number analyzed (Participants) | 12 | 0 | 39 | 0 | 12
months | 14.2 [8.8 to NA] — Upper CI was not reached |  | 16.6 [6.2 to 39.4] |  | 13.6 [8.0 to NA] — Upper CI was not reached

ADVERSE EVENTS:
Arm/Group | Study 2 Arm A | Study 2 Arm B | Study 1 Arm C | Study 3 Arm D | Study 3 Arm E
Serious Adverse Events (participants affected / at risk) | 0/0 | 12/39 | 2/12 | 0/0 | 3/12
Other Adverse Events (participants affected / at risk) | 0/0 | 37/39 | 12/12 | 0/0 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study 2 Arm A (N=0) | Study 2 Arm B (N=39) | Study 1 Arm C (N=12) | Study 3 Arm D (N=0) | Study 3 Arm E (N=12)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
General symptom (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection without neutropenia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study 2 Arm A (N=0) | Study 2 Arm B (N=39) | Study 1 Arm C (N=12) | Study 3 Arm D (N=0) | Study 3 Arm E (N=12)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 13 (82) | 4 (19) | 0 (0) | 2 (29)
Hemoglobin for leukemia studies (Blood and lymphatic system disorders) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 0 (0) | 16 (84) | 2 (8) | 0 (0) | 2 (11)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (6) | 1 (3) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 18 (53) | 3 (14) | 0 (0) | 4 (13)
Diarrhea patients with a colostomy (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (35) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (18) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 7 (10) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 15 (77) | 6 (21) | 0 (0) | 3 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 10 (16) | 3 (5) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 27 (211) | 6 (29) | 0 (0) | 6 (23)
Fever (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
General symptom (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 1 (4) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection without neutropenia (Infections and infestations) | 0 (0) | 7 (10) | 1 (1) | 0 (0) | 0 (0)
Wound-infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase (Investigations) | 0 (0) | 3 (8) | 4 (15) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 13 (34) | 5 (8) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 6 (16) | 0 (0) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 17 (103) | 4 (13) | 0 (0) | 3 (4)
Leukocytes for pediatric BMT studies (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (21)
Neutrophil count decreased (Investigations) | 0 (0) | 17 (84) | 4 (13) | 0 (0) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 15 (97) | 4 (12) | 0 (0) | 3 (5)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 3 (14) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 6 (12) | 1 (1) | 0 (0) | 1 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 18 (45) | 8 (15) | 0 (0) | 4 (31)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 7 (19) | 2 (4) | 0 (0) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 10 (130) | 4 (11) | 0 (0) | 2 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 4 (18) | 0 (0) | 0 (0) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (16) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Cognitive disturbance/learning problems (for pediatrics) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 3 (30) | 2 (7) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (13) | 2 (9) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 2 (9) | 1 (4) | 0 (0) | 0 (0)
Neuropathy - cranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 9 (28) | 4 (9) | 0 (0) | 8 (23)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 12 (31) | 3 (8) | 0 (0) | 3 (21)
Seizure (Nervous system disorders) | 0 (0) | 2 (11) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 6 (18) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (8) | 0 (0) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (9) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (20) | 0 (0) | 0 (0) | 1 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (25) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (32) | 0 (0) | 0 (0) | 2 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 4 (18) | 2 (2) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less